CLINICAL TRIAL: NCT00749086
Title: Prospective Randomized Study of Balloon Kyphoplasty and Vertebroplasty in Subacute (Older Than 6 Weeks) Osteoporotic Vertebral Fractures (STIC2)
Brief Title: Comparison of Balloon Kyphoplasty and Vertebroplasty in Subacute Osteoporotic Vertebral Fractures
Acronym: OSTEO+6
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060108
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Osteoporotic Vertebral Fracture; Between T5 and L5; Chronic Arthritis, Longer Than Six Weeks Duration
Keywords: Osteoporosis; Non-traumatic vertebral fracture; Vertebral compression; Balloon kyphoplasty; Vertebroplasty
MeSH Terms: conditions — Osteoporosis | interventions — Kyphoplasty; Vertebroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): balloon kyphoplasty
  Interventions: Device: balloon kyphoplasty
- 1 (Active Comparator): vertebroplasty
  Interventions: Procedure: vertebroplasty

INTERVENTIONS:
Device: balloon kyphoplasty — Balloon Kyphoplasty, a variant of Vertebroplasty, in which a balloon is first placed into the fractured vertebra and inflated with fluid in order to create a cavity. Then, the balloon are deflated and removed. This may restore part of the vertebral height loss due to the fracture and facilitate the injection of the cement with low pressure.
  Arms: 2
Procedure: vertebroplasty — Vertebroplasty consisting in the percutaneous injection into the fractured vertebra of polymethylmetacrylate cement (the cement used to fix prosthesis in joint replacement) through a posterior route through the vertebral pedicles under radiological guidance
  Arms: 1

SUMMARY:
This study aims to compare two treatments in subacute (more than 6 week duration) non-traumatic (usually osteoporotic) vertebral fractures. The two treatments are the following:

1. Vertebroplasty consisting in the percutaneous injection into the fractured vertebra of polymethylmetacrylate cement (the cement used to fix prosthesis in joint replacement) through a posterior route through the vertebral pedicles under radiological guidance.
2. Balloon Kyphoplasty which consists of placing through a percutaneous posterior approach under radiological guidance, into the fractured vertebra a balloon which is inflated with fluid and creates a cavity. This may restore part of the vertebral height loss due to the fracture. In addition, after balloon deflation, polymethylmetacrylate cement is injected with low pressure into the created cavity to fix fracture reduction. The study will indicate if balloon kyphoplasty is able to restore vertebral height of the fractured vertebra better than vertebroplasty.

DETAILED DESCRIPTION:
Vertebral compression fractures can occur at any level in the vertebral column but the most frequent ones occur at the thoracic (T8-T12) and lumbar spine (L1 and L4). Multiple vertebrae are often concerned. Vertebral fractures are characterized by height reduction of the involved vertebral bodies and very often also by kyphosis and laterally dorsal pain laterally irradiating towards the two sides of the back. A spontaneous improvement of this pain can occur spontaneously within 6 to 12 weeks, but a large number of patients develop a chronic pain and associated morbidity, due to the side effects caused by the fractureThe main cause (85%) of non-traumatic vertebral compression fractures is osteoporosis, in particular in elderly patients. In osteoporotic vertebral fractures older than 6 weeks, conservative management is purely symptomatic, with no effect on the compression fracture itself. Two alternatives are available: Percutaneous Vertebroplasty and Percutaneous Balloon Kyphoplasty

1. Percutaneous Vertebroplasty is a percutaneous treatment of vertebral fractures which is used now for more than 25 years. It was first reported in aggressive vertebral hemangiomas and vertebral malignancies and than in osteoporotic vertebral fractures. More recently, vertebroplasty was used in traumatic vertebral fracture.Vertebroplasty is performed under fluoroscopic guidance with the patient in prone position under general or local anesthesia and conscious sedation. A trocar needle is inserted through a posterior approach into the vertebral neural arch and pedicle, up to the fractured vertebral body. Depending on cases a unilateral or bilateral approach is used. A bilateral approach is used in the cases of traumatic fractures. Once the needle is well positioned into the vertebral body as checked on apical and Lateral views, a radio-opaque cement, in a viscous phase, is slowly injected into the vertebral body under continuous fluoroscopic control. The injection is stopped in case of cement leakage outside from the vertebral body. Polymethylmetacrylate is the most commonly used cement. Its biologic compatibility is well established since used in orthopedic surgery for many decades. Some operators are reluctant to use a non-resorbable cement in young patients. However, to date, the ideal resorbable injectable cement to be discovered. Vertebroplasty allows rapid fracture fixation and decrease in pain, thus allowing the patient to resume walking and daily activities in the days following the procedure. Vertebroplasty does not reduce significantly the kyphosis angle due to the fracture unless nonunion is present in the fracture line.
2. Percutaneous Balloon Kyphoplasty is a variant of vertebroplasty which is performed under general anaesthesia using the KyphX® System (Medtronic, Sunnyvale, California). Balloon kyphoplasty aims at restore vertebral height of the fractured vertebra using an inflatable balloon prior to inject surgical cement (PMMA) into the vertebral body and fix the fracture. It is an expensive technique costing around 4,000 euros for up to 2 vertebrae in the same patient. The surgical technique for the procedure has been described by Lieberman et al. A bilateral approach is chosen to insert working cannulas into the posterior part of the vertebral body. Fluoroscopy is used to insert the tools and control the procedure. With reaming tools, two working channels are created and the balloons are inserted. The balloons are available in lengths of 10, 15 and 20 mm.The two balloons(one on each side) should ideally be centered at middle height between the superior and inferior endplates and in the anterior two-thirds of the vertebral body. Balloon placement into the vertebral body is checked using radiopaque markers at the two extremities of the balloon. Once inserted, the balloons are inflated using visual, volume and pressure control to create a cavity. Inflation is stopped when one of the following inflation endpoints is reached: pressure raised over 400 psi, balloon contacts one of the cortical bone of the vertebra or reaching maximal balloon inflation volume. The balloons are then deflated and removed. The mean balloon inflation volume is 2 to 3ml. The Bone Filler Device, filled before with 1.5 ml of polymethylmethacrylate (PMMA), is then advanced through the working cannula towards the anterior part of the cavity and cement is slowly extruded by a stainless steel stylet, acting as a plunger. When the amount of cement from the first Bone Filler Device is delivered in the cavity, it is removed and another Bone Filler Device is advanced through the working cannula. This step is repeated till a complete fill of the cavity is obtained. The same procedure is repeated through the other working cannula at the contra-lateral pedicle. Filling of the cavity with highly viscous PMMA is performed under continuous fluoroscopic control.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to undergo the vertebroplasty or Balloon kyphoplasty procedure
* Patient has read and sign the informed consent
* Male or female, 50 years or older
* One or two non-traumatic vertebral fracture(s):

  * Of osteoporotic origin (low speed trauma such as fall from his own height or less than 80 cm)
  * Fracture(s) older than 6 weeks duration after the onset of pain related to the fracture· The fracture(s) exhibit(s) high signal intensity on T2-weighted images and a benign appearance at MRI
* Persistent pain despite medical treatment according to VAS ≥ 5 or a last resort to morphine treatment
* The patient will be able to receive the selected protocol treatment within 15 days after treatment randomization.
* The benign nature of the vertebral fracture has to be confirmed by the results of the biopsy performed during vertebroplasty or balloon kyphoplasty.

Exclusion Criteria:

* Patient with a vertebral fracture of less than 6 week duration after onset of fracture-related symptoms.
* Neurological signs related to the vertebral fracture to treat
* History of surgical or percutaneous spine treatment except simple discectomy at a single or multiple vertebral levels with no residual pain.
* Patient with more than 2 fractures corresponding to the inclusion criteria (old fractures are not taken into account)
* Known allergy to a contrast media or to one of the cement components used for kyphoplasty.
* More than two recent vertebral fractures
* Current infection
* Impossibility to perform the percutaneous approach of the vertebra to treat.
* Known allergy to a contrast media or to one of the cement components used for kyphoplasty.
* Reduction by more than 50% of the anteroposterior width of the bony spinal canal due to the vertebral fracture to treat.
* Vertebral fracture with loss of 90%or more of the vertebral body height
* Malignant and traumatic vertebral fractures
* Contraindication to MRI :

  * Metallic implant : pace-maker, no auditive implant , metallic vascular or movable cardiac device
  * Metallic surgical clips Claustrophobia
* Evolutive cardiac disease nonreactive to medical treatment
* Patient presenting a non correctable spontaneous or therapeutic coagulation disorder.
* Presence of an unexplained biological inflammatory syndrome with VS≥20
* Non compliant patient: Impossibility to participate to the study and to be followed up for 1 year.
* Pregnant or breast feeding women
* Patient not affiliated to social security

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2007-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Modification of the kyphotic angle of every treated vertebra (between the preoperative angle and measured after 1 year follow-up) | 1 year

SECONDARY OUTCOMES:
Evaluation of pain through the visual analog scale | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Functional scale (EIFEL) for lumbar pain | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Evaluation of quality of life (QUALEFFO - Short Form SF12) | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Analgesics intake according to the WHO classification (Classes 1, 2 and 3). | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Evaluation of kyphotic angle and global thoracic and lumbar angulations | At each follow-up visit (J-20 to J-7 - J6 - J45 - J90 - J180 - J360) :
Measurement of anterior, median and posterior height of the discs adjacent to the fracture; | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Measurement of disc angles adjacent to the fracture; | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Number of new vertebral fractures documented radiologically | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Medico-economic follow-up on 10% of the randomly selected patients:o Cost of intervention.o Cost of prescribed medicines.o Cost of follow-up visits.o Cost of subsequent hospitalization.o Cost of complications. | J-20 to J-7 - J6 - J45 - J90 - J180 - J360
Follow-up of anterior, median and posterior height of the treated vertebral body, obtained by making an average of all measurements, on 3 cuts CT-SCAN on the sagittal level : lateral right, median and lateral left | preoperative, at J6 and at J360
Intensity of signal with T2 sequence | preoperative and at J360

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Denis LAREDO, M.D.,PR., Principal Investigator — AP-HP Assistance Publique- Hôpitaux de Paris
Locations (1):
- Service de Radiologie, Hôpital Lariboisière, Paris, France